CLINICAL TRIAL: NCT06918171
Title: Clinical Efficacy of Open Reduction and Suture Bridge Fixation for PCL Tibial Avulsion Fractures
Acronym: fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-HG-2025-035
Record Dates: First submitted 2025-03-29; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Tibial Plateau Fracture
Keywords: fracture fixation; Retrospective study
MeSH Terms: conditions — Tibial Plateau Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Efficacy of Open Reduction and Anchor Suture Bridge Fixation (Experimental): Under general anesthesia, patients were positioned prone, and a midline posterior incision was made at the level of the popliteal fossa. After incising the fascia, careful dissection was undertaken to expose the posterior joint capsule and fracture fragment, with particular attention to safeguarding the neurovascular structures. Once the fracture site was fully exposed, hematoma and any interposing soft tissue were meticulously cleared to prepare for reduction. The avulsed bone fragment, located at the PCL insertion site, was identified and prepared for fixation. A suture anchor (Johnson & Johnson, USA) was carefully implanted into the prepared osseous bed. The suture threads were passed anteriorly around the PCL and configured in a figure-of-eight pattern to achieve precise anatomical reduction of the fracture fragment. To enhance fixation stability, two extracortical anchors (Johnson & Johnson, USA) were additionally positioned approximately 2 cm distal to the fracture site, securin
  Interventions: Procedure: Clinical Efficacy of Open Reduction and Anchor Suture Bridge Fixation

INTERVENTIONS:
Procedure: Clinical Efficacy of Open Reduction and Anchor Suture Bridge Fixation — Under general anesthesia, patients were positioned prone, and a midline posterior incision was made at the level of the popliteal fossa. After incising the fascia, careful dissection was undertaken to expose the posterior joint capsule and fracture fragment, with particular attention to safeguarding the neurovascular structures. Once the fracture site was fully exposed, hematoma and any interposing soft tissue were meticulously cleared to prepare for reduction. The avulsed bone fragment, located at the PCL insertion site, was identified and prepared for fixation. A suture anchor (Johnson & Johnson, USA) was carefully implanted into the prepared osseous bed. The suture threads were passed anteriorly around the PCL and configured in a figure-of-eight pattern to achieve precise anatomical reduction of the fracture fragment. To enhance fixation stability, two extracortical anchors (Johnson & Johnson, USA) were additionally positioned approximately 2 cm distal to the fracture site, securing

SUMMARY:
Abstract Background: Posterior cruciate ligament (PCL) tibial avulsion fractures significantly impair knee function; however, optimal surgical fixation approaches are not agreed upon. The investigators performed this study to compare the clinical outcomes of PCL tibial avulsion fractures treated with open reduction and anchor suture bridge fixation.

Methods: A total of 17 patients underwent open reduction and anchor suture bridge fixation following injury. The investigators recorded operation time, intraoperative and postoperative complications, and used imaging to assess fracture reduction and healing. Visual Analog Scale (VAS), Lysholm Knee Scoring Scale, International Knee Documentation Committee (IKDC) score, and knee range of motion (ROM) were evaluated preoperatively, 3 months postoperatively, and at final follow-up.

DETAILED DESCRIPTION:
Patient Selection This study was approved by the Ethics Committee of the Second Affiliated Hospital of Soochow University. The ethics number was: JD-HG-2025-035. From January 2019 to December 2023, patients diagnosed with PCL tibial avulsion fractures and treated with open reduction combined with anchor fixation at our center were evaluated for inclusion. Inclusion criteria were: (1) a clear diagnosis of PCL tibial avulsion fracture verified through preoperative radiographs and computed tomography (CT), with classification as type II or III based on the Griffith system (a modified Meyers and McKeever scale)[16]; (2) patients aged 18 years or older; (3) surgical management within two weeks post-injury; and (4) absence of additional ligament or meniscal injuries in the affected knee. Exclusion criteria were: (1) concurrent ligament or meniscal injuries confirmed via magnetic resonance imaging (MRI); (2) prior surgical procedures or traumatic injuries involving the same knee; (3) severe systemic diseases that could interfere with surgical outcomes; and (4) insufficient clinical or radiographic follow-up data. In total, 17 patients (9 males and 8 females), with an average age of 49 ± 12 years, who satisfied all inclusion and exclusion criteria, were ultimately included for analysis.

Surgical Techniques All surgeries were carried out by the same experienced orthopedic surgeon to ensure procedural consistency. Under general anesthesia, patients were positioned prone, and a midline posterior incision was made at the level of the popliteal fossa. After incising the fascia, careful dissection was undertaken to expose the posterior joint capsule and fracture fragment, with particular attention to safeguarding the neurovascular structures. Once the fracture site was fully exposed, hematoma and any interposing soft tissue were meticulously cleared to prepare for reduction. The avulsed bone fragment, located at the PCL insertion site, was identified and prepared for fixation. A suture anchor (Johnson & Johnson, USA) was carefully implanted into the prepared osseous bed. The suture threads were passed anteriorly around the PCL and configured in a figure-of-eight pattern to achieve precise anatomical reduction of the fracture fragment. To enhance fixation stability, two extracortical anchors (Johnson & Johnson, USA) were additionally positioned approximately 2 cm distal to the fracture site, securing the suture construct effectively. Intraoperative fluoroscopy was utilized to verify proper fracture reduction and secure fixation. Upon confirmation, the surgical site was irrigated, hemostasis was achieved, and the incision was closed in layers.

Postoperative Management Postoperatively, all patients were immobilized with a hinged knee brace locked in full extension for the initial 2 weeks, and partial weight-bearing with crutches was permitted as tolerated. Passive knee range-of-motion exercises (0°-60°) were initiated under supervised rehabilitation 2 weeks after surgery. At 4-6 weeks postoperatively, progressive weight-bearing was encouraged according to fracture healing confirmed by radiographic assessment, and knee flexion was gradually increased (0°-90°). After 8 weeks, patients transitioned to full weight-bearing, and active muscle strengthening and proprioception training programs were initiated.

Clinical Assessments Clinical outcomes were comprehensively assessed at three distinct time points: prior to surgery, at 3 months postoperatively, and at the final follow-up visit. The key evaluation parameters included pain intensity, knee joint function, range of motion (ROM), fracture healing, and postoperative complications. Pain severity was quantified using the Visual Analog Scale (VAS; 0-10 points), where 0 indicates no pain and 10 represents the worst possible pain. Functional outcomes were evaluated with two well-established scoring systems: the Lysholm Knee Scoring Scale (ranging from 0 to 100, where higher scores indicate better knee function) and the International Knee Documentation Committee (IKDC) subjective knee assessment (also ranging from 0 to 100, with higher values reflecting superior functional status). Knee ROM, encompassing both maximal flexion and extension, was measured using a standard goniometer. Fracture union was assessed via routine anteroposterior and lateral radiographs, with successful healing defined as the presence of continuous cortical alignment and trabecular bridging at the fracture site, without detectable fracture lines. In addition, any postoperative complications, including infection, neurovascular injuries, hardware-related issues, implant discomfort, or the necessity for reoperation, were meticulously documented during each follow-up assessment.

Statistical Analysis Statistical analyses were conducted using SPSS software (version 26.0). Continuous variables were expressed as mean ± standard deviation (SD) or as median with interquartile range (IQR), depending on the data distribution. The Shapiro-Wilk test was applied to examine the normality of continuous variables. Comparisons of clinical outcomes, including VAS pain scores, Lysholm knee scores, IKDC scores, and knee range of motion (ROM), across preoperative and postoperative time points were evaluated using the Friedman test for repeated measures, with Wilcoxon signed-rank tests employed for post hoc pairwise comparisons. Categorical variables, such as complication rates, were summarized as frequencies and percentages. A P-value < 0.05 was considered indicative of statistical significance in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* A clear diagnosis of posterior cruciate ligament (PCL) tibial avulsion fracture, verified through preoperative radiographs and computed tomography (CT), with classification as type II or III based on the Griffith system (a modified Meyers and McKeever scale).
* Patients aged 18 years or older.
* Surgical management within two weeks post-injury.
* Absence of additional ligament or meniscal injuries in the affected knee, confirmed via magnetic resonance imaging (MRI).

Exclusion Criteria:

* Concurrent ligament or meniscal injuries in the affected knee, confirmed via MRI.
* Prior surgical procedures or traumatic injuries involving the same knee.
* Severe systemic diseases that could interfere with surgical outcomes (e.g., uncontrolled diabetes, severe cardiovascular disease).
* Insufficient clinical or radiographic follow-up data.

Additional Information:

In total, 17 patients (9 males and 8 females), with an average age of 49 ± 12 years, who satisfied all inclusion and exclusion criteria, were ultimately included for analysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Score | 6 months after surgery
  The Visual Analog Scale (VAS) Score is used to assess the intensity of pain experienced by patients. The VAS is a continuous scale comprising a 100-mm line, where the minimum value is 0 (representing no pain) and the maximum value is 10 (representing the worst imaginable pain). A higher score indicates a worse outcome, reflecting greater pain intensity. The mean VAS score across all participants will be reported to evaluate the average pain level at 6 months post-surgery.
Lysholm Knee Scoring Scale | 6 months after surgery
  The Lysholm Knee Scoring Scale is used to evaluate knee function and symptoms. The scale ranges from a minimum value of 0 to a maximum value of 100. A higher score indicates a better outcome, reflecting improved knee function and fewer symptoms. The scale assesses factors such as pain, instability, locking, swelling, and the ability to perform activities like climbing stairs or squatting. The mean Lysholm score across all participants will be reported to evaluate the average knee function at 6 months post-surgery.
International Knee Documentation Committee Score | 6 months after surgery
  The International Knee Documentation Committee (IKDC) Score is used to evaluate knee function, symptoms, and the ability to engage in sports activities following surgery. The IKDC Score ranges from a minimum value of 0 to a maximum value of 100. A higher score indicates a better outcome, reflecting improved knee function, fewer symptoms, and better overall knee health. The score assesses aspects such as pain, swelling, knee stability, and the ability to perform daily activities and sports. The mean IKDC score across all participants will be reported to evaluate the average knee function and sports activity level at 6 months post-surgery.
Range of Motion | 6 months after surgery
  The Range of Motion (ROM) of the knee is measured to assess the degree of knee flexion and extension following surgery. ROM is evaluated using a goniometer, with measurements recorded in degrees. The minimum value for knee flexion is 0 degrees (indicating no flexion, i.e., a fully extended knee), and the maximum value can reach up to approximately 135 degrees in a healthy knee (indicating full flexion). For extension, the minimum value is 0 degrees (full extension), while negative values (e.g., -5 degrees) may indicate an extension deficit. A greater ROM, particularly in flexion, indicates a better outcome, reflecting improved knee mobility and function. The mean flexion and extension angles across all participants will be reported to evaluate the average knee mobility at 6 months post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The medical record system and imaging system of the Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes